CLINICAL TRIAL: NCT00337532
Title: A Phase II Trial Neoadjuvant Paclitaxel and Cisplatin in Patients With Locally Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-384
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2008-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Paclitaxel; Cisplatin

ARMS (1):
- paclitaxel-cisplatin combination regimen (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: cisplatin

INTERVENTIONS:
Drug: Paclitaxel — Sterile solution mixed with 0.9% saline or 5% glucose solution 500mL, 3-hour Continuous infusion, Level 0: 175 mg/m2, Level 1: 140 mg/m2, Level 2: 105 mg/m2 (dose reduction in function of toxicity), Day 1 of each cycle, max of 3 cycles; each cycle of 21 days ± 3 days.
Drug: cisplatin — solution mixed with 0.9% saline 500mL, 30 to 90 min intravenous infusion, Level 0: 75 mg/m2, Level 1: 60 mg/m2, Level 2: 45 mg/m2 (dose reduction in function of toxicity), Day 1 of each cycle, max of 3 cycles; each cycle of 21 days ± 3 days.

SUMMARY:
The purpose of this clinical research study is to learn if a paclitaxel-cisplatin combination regimen given in the neoadjuvant setting is active in locally advanced head and neck cancer. the safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, Stage II-IV (except M1), hand and neck cancer
* > = 1 measurable lesion
* not been previously treated for head and neck cancer

Exclusion Criteria:

* history of another malignancy
* organ allografts
* pre-exiting neuropathy > = CTC grade 2

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Tumor response rate of locally advanced head and neck cancer to a paclitaxel-cisplatin combination regimen in a neoadjuvant setting and administered during maximum 3 cycles.

SECONDARY OUTCOMES:
Toxicity for maximum 3 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- South Korea (2):
  - Local Insitution, Seoul
  - Local Institution, Seoul